CLINICAL TRIAL: NCT04264520
Title: Initial Intervention Efficacy for an Online PTSD Intervention for Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed institutions and was no longer able to continue project.
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC Specialized Center of Research Excellence (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00096405
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Perinatal Problems; Post Traumatic Stress Disorder; Post Partum Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Open Label Pilot Trial (no control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTSD Psychoeducation + Skills Intervention (Experimental)
  Interventions: Behavioral: PTSD Psychoeducation + Skills Intervention

INTERVENTIONS:
Behavioral: PTSD Psychoeducation + Skills Intervention — A brief computer-assisted intervention (psychoeducation + skills) for pregnant women with elevated PTSD symptoms.

SUMMARY:
The current study aims to test a brief computer-assisted intervention (psychoeducation + skills) for pregnant women with elevated PTSD symptoms. In this open trial pilot feasibility study, 20 pregnant women in their first trimester will be invited to participate in the study if they endorse elevated PTSD symptoms. Oxytocin and cortisol will be measured at baseline, one month post-intervention, three months post-intervention, and post-delivery to inform the relationship between these hormones, PTSD symptoms, and peripartum/postpartum outcomes. In addition to receiving the psychoeducation + skills intervention during their first trimester, women will be offered a "booster session" intervention following delivery to enhance utilization of skills during a critical period for maternal mental and physical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Fluent in English

Exclusion Criteria:

* Active and severe domestic violence
* Evidence of a significant mental illness or current substance use disorder that would impede the completion of the intervention
* Suicidal individuals deemed at immediate danger or risk (i.e., requiring immediate hospitalization or treatment)
* Women who smoke
* Women who have a metabolic or endocrine disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Intervention for pregnant women, so only women can be included.
Enrollment: 5 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) Total Scores | Baseline to follow-up (follow-up will occur at one-month following the baby's birth)
  The PCL-5 is a 17-item self-report questionnaire designed to assess PTSD symptoms among civilians. In the current study, PCL-5 total scores will be utilized. Specifically, we will examine the impact of the intervention on change in PCL-5 scores across time (i.e., from baseline to post-delivery follow-up). Scores on the PCL-5 range from 0 to 80, with higher scores indicating more symptoms.
Baby's Weight at Birth in Pounds/Ounces | Baseline to birth of baby.
  Each baby's weight (in pounds/ounces) will be derived from the online medical record following delivery. This outcome will be used to determine the relationship between maternal PTSD symptoms (as indexed by the PCL-5 total scores--above) and infant weight at birth.
Total Gestation Length in Weeks | Baseline to birth of baby.
  The total gestation length, in weeks, will be derived from the online medical record following the baby's birth. This outcome will be used to determine the relationship between maternal PTSD symptoms (as indexed by the PCL-5 total scores--above) and total weeks gestation at birth.
Baby's APGAR Score at Birth | Baseline to birth of baby.
  Each baby's APGAR score will be derived from the online medical record following delivery. APGAR scores range from 0-10, with higher scores indicating better health at birth for baby. APGAR scores will be used to determine the relationship between maternal PTSD symptoms (as indexed by the PCL-5 total scores--above) and infant health at birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No